CLINICAL TRIAL: NCT00682240
Title: Morphological and Functional Retinal Changes Following Retinal Photocoagulation Using a Semiautomated Patterned Scanning Laser System in Proliferative Retinopathy or Macular Edema Secondary to Diabetes Mellitus or Retinal Vein Occlusion
Brief Title: Morphological and Functional Retinal Changes Following Retinal Photocoagulation
Acronym: pascal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Katharina Kriechbaum, Ass.Prof.Dr., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Pascal Study
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Proliferative Diabetic Retinopathy; Macular Edema
Keywords: retinal morphology; laser treatment; pascal laser; HD-OCT
MeSH Terms: conditions — Macular Edema

ARMS (4):
- group 3 (Active Comparator): Group 3: 20 patients with proliferative retinopathy secondary to diabetes mellitus or venous occlusion) with need for panretinal photocoagulation.
  Intervention: All patients will receive a multi-session panretinal laser treatment according to the conventional protocol, using a conventional laser system.
  Interventions: Procedure: laser treatment with conventional laser system
- group 2 (Active Comparator): Group 2: 20 patients with proliferative retinopathy secondary to diabetes mellitus or venous occlusion) with need for panretinal photocoagulation randomized into group 2.
  Intervention: This group will receive multi-session panretinal laser treatment. The treatment will be performed using Pascal laser system.
  Interventions: Procedure: laser treatment with PASCAL®
- group 1 (Active Comparator): Group 1: 20 patients with proliferative retinopathy secondary to diabetes mellitus or venous occlusion) with need for panretinal photocoagulation randomized into group1.
  Intervention: One group will receive a single-session panretinal laser treatment, performed using Pascal laser system.
  Interventions: Procedure: laser treatment with PASCAL®
- group 4 (Active Comparator): Group 4: 20 patients with persistent central or para-central diabetic macular edema receiving focal or grid laser treatment. As the treatment will be performed according to the conventional protocol (single spot), only the Pascal laser system will be used.
  Intervention: focal or grid laser treatment
  Interventions: Procedure: laser treatment with PASCAL®

INTERVENTIONS:
Procedure: laser treatment with PASCAL® — panretinal laser treatment - single-session
  Other Names: PASCAL® (Pattern Scan Laser, OptiMedica ® Corporation)
  Arms: group 1
Procedure: laser treatment with PASCAL® — panretinal laser treatment - multi-session
  Other Names: The PASCAL® (Pattern Scan Laser, OptiMedica ® Corporation)
  Arms: group 2
Procedure: laser treatment with PASCAL® — grid / focal laser treatment
  Other Names: PASCAL® (Pattern Scan Laser, OptiMedica ® Corporation)
  Arms: group 4
Procedure: laser treatment with conventional laser system — panretinal laser treatment - multi-session according to the conventional protocol, using a conventional laser system
  Arms: group 3

SUMMARY:
Imaging of retinal morphological changes with time secondary to laser treatment as assessed with high definition optical coherence tomography (OCT). Furthermore changes in retinal function as an effect of treatment will be documented by visual acuity testing using ETDRS charts and microperimetry. The change in vascular leakage will be assessed by performing fluorescein angiography, flare counts will be performed monthly.

DETAILED DESCRIPTION:
Hypertension and diabetes are widespread diseases in our modern society and due to the comfortable, but often unhealthy "western world" lifestyle, the population suffering from its consequences is constantly growing. Vascular pathologies affect the body's entire vascular system subsequently including the circulation and vessels in the eye. For these reasons, after diabetic retinopathy and vein occlusions rank among the most common vascular disorders of the retina, with the highest incidence in a population over the age of 60. As to prevent severe vision loss due to complications induced by these angiopathies, panretinal or segmental laser coagulation is recommended as standard treatment of proliferative retinopathy. So far patients who undergo panretinal coagulation typically receive between 1200 and 1500 lasers spots in two to four sessions over the course of 2 to 4 weeks. Clinical guidelines recommend not exceeding the number of more than 900 applied laser spots per session, due to the development of possible reversible exudative reaction e.g. macular edema. However, the performance of a panretinal photocoagulation is so far a time consuming procedure which is generally painful for the patient. For these reasons new laser systems were developed aiming to solve these obvious drawbacks. Main improvement of these systems is the reduction of the laser burn durations per spot and to enable therefore the rapid application of a large number of spots in a preset pattern. Treatment with reduced pulse duration is associated with less pain for the patient and, compared to several sessions requiring about 30 minutes each when using a conventional laser system, treatment time for a complete panretinal treatment could be significantly reduced. The PASCAL® Laser (Pattern Scan Laser, OptiMedica® Corporation, Santa Clara, CA, USA) is a new commercially available laser system confirming all these requirements.

As the first study part (group I and II) we propose a controlled randomized comparison of single session to conventional multisession panretinal laser treatment, using the Pascal laser system for the single-session protocol and the Pascal laser system or the conventional laser system for the multi-session protocol. Development and regression of a retinal exudative reaction and the eventual onset of transient macular edema will be observed and documented. The morphological changes within the retina induced by laser burns will be imaged mainly using optical coherence tomography techniques. In regard to determine the lowest laser intensity as possible to produce a visible morphologic effect within small retinal areas different laser intensities will be used for photocoagulation of retinal segments to show the effect of a "sub-threshold" and gentle laser burn.

As a second study part (group III), grid pattern laser coagulation will be performed in a conventional way using the Pascal laser system. In a small area of the retinal perifoveal zone showing macular edema, morphologic effects of photocoagulation using titrated low, sub threshold or threshold laser energy will be analyzed using OCT.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 18 years
* Patients with either retinopathy/maculopathy secondary to diabetes mellitus type I or II with medical indication for segmental or panretinal laser coagulation or with necessity for completion of previous incomplete laser photocoagulation.
* Patients with proliferative diabetic retinopathy requiring panretinal laser treatment (Group 1, 2 and 3)
* Patients with macular edema requiring central focal or grid laser treatment (Group 4).

Exclusion criteria:

* A condition that would preclude a patient for participation in the study in opinion of investigator, e.g., unstable medical status including glycemic control and blood pressure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Retinal morphological changes with time secondary to laser treatment as assessed with optical coherence tomography (OCT). | 2007-2014

SECONDARY OUTCOMES:
changes in retinal function as an effect of treatment, documented by visual acuity testing and microperimetry. The change in vascular leakage will be assessed by performing fluorescein angiography, flare counts will be performed monthly. | 2007-2009

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Schmidt-Erfurth, MD, Study Chair — Medial University of Vienna, Dept. of Ophthalmology; Katharina Kriechbaum, MD, Principal Investigator — Medical University of Vienna; Matthias Bolz, MD, Principal Investigator — Medical University of Vienna; Sonja Prager, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Dept. of Opthalmology, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Deak GG, Bolz M, Prager S, Ritter M, Kriechbaum K, Scholda C, Schmidt-Erfurth U; Diabetic Retinopathy Research Group Vienna. Photoreceptor layer regeneration is detectable in the human retina imaged by SD-OCT after laser treatment using subthreshold laser power. Invest Ophthalmol Vis Sci. 2012 Oct 9;53(11):7019-25. doi: 10.1167/iovs.12-10196. Print 2012 Oct. PMID 22956609